CLINICAL TRIAL: NCT07191236
Title: Telemonitoring for High-risk Pregnancies in an International Context (PregnaDigit EU): a Hybrid Type 2 Study
Brief Title: Development of an International Remote Digital Care System for Accessible, Inclusive and Sustainable Pregnancy Care
Acronym: PregnaDigit EU
Status: Enrolling by invitation | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Mireille Bekker, Prof. Dr., UMC Utrecht
Other Study IDs: OBS_24U-1738; 240036 (Other Grant/Funding Number: EIT Health)
Record Dates: First submitted 2025-09-03; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Telemedicine; Digital Health; Pregnancy Complications
Keywords: Telemedicine; Digital Health; Pregnancy; Pregnant People; Pregnancy Complications; Implementation science
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Telemonitoring cohort: This prospective cohort consists of pregnant individuals with high-risk complications who require frequent cardiotocography (CTG) monitoring according to local protocol. Instead of receiving in-hospital CTG monitoring, participants will perform CTG recordings at home, with optional blood pressure (BP) measurements. Recordings are transmitted securely and reviewed by trained obstetric healthcare providers, followed by telephone or video contact. This cohort represents real-world implementation of remote digital pregnancy care and enables evaluation of clinical and implementation outcomes.

SUMMARY:
Pregnancy care is under increasing pressure due to a rising number of women needing medical care, a shortage of obstetric healthcare professionals, and growing healthcare costs. For women with high-risk pregnancies, this often leads to frequent hospital visits or admissions for monitoring, which can be stressful and time consuming. Remote digital care offers a promising alternative by allowing pregnant individuals to perform monitoring from home while remaining under medical supervision.

This study will evaluate the use of telemonitoring in pregnancy care in four European hospitals. Participants with high-risk pregnancies who require frequent cardiotocography (CTG) monitoring and blood pressure (BP) measurements will use certified home devices to record fetal and maternal health data. Instead of hospital-based monitoring, CTG and BP measurements will be performed at home and assessed by trained healthcare professionals.

The main purpose of the study is to investigate whether home monitoring is a safe and acceptable alternative to in-hospital monitoring, and to identify what is needed for successful national and international implementation of remote digital pregnancy care. The investigators will collect clinical and implementation outcomes. By doing so, this study aims to keep pregnancy care accessible for all women, improve patient well-being, and reduce pressure on the healthcare system.

DETAILED DESCRIPTION:
This study investigates the implementation and effectiveness of telemonitoring using cardiotocography (CTG) and blood pressure (BP) home monitoring in four European academic hospitals. RDPC allows pregnant individuals with high-risk complications to conduct CTG recordings at home, which are then reviewed by trained obstetric healthcare providers through secure digital platforms. This approach has the potential to replace hospital-based monitoring, reduce healthcare consumption, and improve patient well-being while maintaining safety.

The study is conducted in four tertiary referral centers for obstetric care: University Medical Center Utrecht and Erasmus Medical Center in the Netherlands, Vall d'Hebron University Hospital in Spain, and Karolinska University Hospital in Sweden. These hospitals serve large and diverse populations and have extensive experience with managing high-risk pregnancies, providing an international perspective on the implementation and effectiveness of RDPC.

Telemonitoring will be conducted with CE-certified CTG devices (PregnaBit Pro with PregnaOne Platform or Mosos CTG by ICT/HCTS, or the Nemo fetal monitoring system by Nemo Healthcare), and in some centers, blood pressure will be monitored using Microlife WatchBP devices. All devices are CE-certified and not classified as investigational products in this study.

The study follows a hybrid type 2 implementation-effectiveness design. First, this study will assess clinical outcomes of participants undergoing telemonitoring. The study will investigate adverse maternal and perinatal outcomes to ensure that home monitoring is a safe alternative to hospital-based care. To further assess the clinical effectiveness of telemonitoring, investigators will evaluate health care consumption of pregnant participants during telemonitoring, such as the number of days each participant received telemonitoring and number and indications of unplanned hospital visits and admissions. These data will provide insight into the health care demands associated with the telemonitoring care pathways. These measures will provide valuable insights into the efficiency and scalability of telemonitoring.

In addition to clinical outcomes, this study will evaluate implementation outcomes across three sequential phases: pre-implementation, implementation, and post-implementation. Outcomes are based on the taxonomy of Proctor et al., including acceptability, adoption, appropriateness, feasibility, fidelity, costs, penetration, and sustainability. Implementation data will be collected from patients and obstetric healthcare professionals, and hospital systems through questionnaires, interviews, and structured data analyses.

Data will be collected and managed in Castor EDC, a GCP-classified web-based data management platform. Data entry will be performed by local research teams, with centralized oversight and quality assurance procedures. Analyses will include descriptive statistics, logistic regression to evaluate the composite clinical endpoint, and regression models to identify factors influencing implementation success.

Ultimately, this study aims to generate knowledge, recommendations, and scalable care models that enable sustainable nationwide and international integration of remote digital pregnancy care, keeping care accessible while reducing system pressure and costs.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* A singleton pregnancy of ≥26+0 weeks of gestation (UMCU, EMC, and Vall d'Hebron) or ≥24+0 weeks of gestation (Karolinska)
* Able to give informed consent.
* Proficiency in English or the local language (Dutch, Spanish or Swedish)
* The presence of a complication requiring CTG monitoring according to local protocol

Exclusion Criteria:

* Pregnancy complications requiring intravenous (IV) anti-hypertensive therapy
* Expected obstetric intervention within 48 hours
* Current blood pressure ≥160 mmHg systolic or ≥110 mmHg diastolic
* Active antepartum hemorrhage
* CTG abnormalities suggestive of fetal stress or hypoxia
* Residence located more than a 30-minute drive from any hospital (not necessarily the hospital initiating home monitoring)
* Presence of an implanted medical device (e.g. pacemaker)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at four European university hospitals: University Medical Center Utrecht (UMCU) (Netherlands), Erasmus Medical Center (EMC) Rotterdam (Netherlands), Vall d'Hebron University Hospital (Spain), and Karolinska University Hospital (Sweden). The study population consists of pregnant individuals receiving care for high-risk pregnancies that require frequent cardiotocography (CTG) monitoring according to local clinical protocols. Instead of hospital-based monitoring, eligible participants will perform CTG recordings from home using telemonitoring systems.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome: composite of adverse perinatal and maternal events | During pregnancy up to six months postpartum
  The primary clinical outcome is a composite measure of adverse perinatal and maternal events. This dichotomous composite is defined as the occurrence of one or more of the following:
  * Perinatal mortality (maternal, fetal, or neonatal)
  * Low neonatal condition at birth: 5-minute Apgar score < 7 and/or arterial cord blood pH < 7.05
  * Maternal morbidity, including one or more of:
  Hypertensive crisis requiring intravenous antihypertensive medication and/or MgSO4 for eclampsia prevention Eclampsia (new-onset, generalized tonic-clonic seizures or coma in a woman with preeclampsia) HELLP syndrome (hemolysis, elevated liver enzymes, and low platelet count) Venous thromboembolism (deep vein thrombosis or pulmonary embolism) Maternal admission to an Intensive Care Unit (ICU) Admission of the newborn to a Neonatal Intensive Care Unit (NICU) ≥ 24 hours
  -Caesarean section.
Implementation outcome: Proctor Acceptability | Questionnaire obstetric health care providers: at baseline and at the end of the implementation phase. Questionnaire pregnant participants: 5 days after starting telemonitoring. Depending on each site and participant questionnaires are send out in 2025.
  Implementation outcomes will be analyzed according to the taxonomy of Proctor et al. Proctor defined eight implementation outcomes: acceptability, adoption, appropriateness, feasibility, fidelity, costs, penetration and sustainability.
  Acceptability: The perception that telemonitoring is agreeable, palatable or satisfactory among obstetric healthcare providers and pregnant participants. Assessment method is by questionnaires.
Implementation outcome: Proctor Adoption | Qualitative analysis of semi-structures interviews: pre-implementation phase (dec-jan 2025)Questionnaire obstetric health care providers: at baseline and at the end of the implementation phase (2025).
  Implementation outcomes will be analyzed according to the taxonomy of Proctor et al. Proctor defined eight implementation outcomes: acceptability, adoption, appropriateness, feasibility, fidelity, costs, penetration and sustainability.
  Adoption: The intention to start telemonitoring among obstetric healthcare providers. Assessment method: qualitative analysis of semi-structured interviews and questionnaire.
Implementation outcome: Proctor Appropriateness | Questionnaire obstetric health care providers: at baseline and at the end of the implementation phase. Depending on each site and participant questionnaires are send out in 2025.
  Implementation outcomes will be analyzed according to the taxonomy of Proctor et al. Proctor defined eight implementation outcomes: acceptability, adoption, appropriateness, feasibility, fidelity, costs, penetration and sustainability.
  Appropriateness: The perceived fit, relevance, or compatibility of telemonitoring among obstetric healthcare providers and pregnant participants.. Assessment method: questionnaire.
Implementation outcome: Proctor Costs | Whole study duration up untill the end of data analysis Feb 2028
  Implementation outcomes will be analyzed according to the taxonomy of Proctor et al. Proctor defined eight implementation outcomes: acceptability, adoption, appropriateness, feasibility, fidelity, costs, penetration and sustainability.
  Costs: The cost impact analysis of telemonitoring. Assessment method: Metro Maps and Time Driven Activity Based Costing (TDABC)
Implementation outcome: Proctor Feasibility | Questionnaire obstetric health care providers: at baseline and at the end of the implementation phase. Depending on each site and participant questionnaires are send out in 2025.
  Implementation outcomes will be analyzed according to the taxonomy of Proctor et al. Proctor defined eight implementation outcomes: acceptability, adoption, appropriateness, feasibility, fidelity, costs, penetration and sustainability.
  Feasibility: The extent to which telemonitoring can be successfully used or carried out within the hospital by obstetric healthcare providers. Assessment method is by questionnaires.
Implementation outcome: Proctor Fidelity | Whole study duration up untill the end of data analysis Feb 2028
  Implementation outcomes will be analyzed according to the taxonomy of Proctor et al. Proctor defined eight implementation outcomes: acceptability, adoption, appropriateness, feasibility, fidelity, costs, penetration and sustainability.
  Fidelity: The extent to which telemonitoring is implemented as it was described in the original protocol. Assessment method: Number of wrongful inclusions, eligbile patients missed, adherence to the predefined protocol.
Implementation outcome: Proctor Penetration | Questionnaire obstetric health care providers: at baseline and at the end of the implementation phase. Depending on each site and participant questionnaires are send out in 2025.
  Implementation outcomes will be analyzed according to the taxonomy of Proctor et al. Proctor defined eight implementation outcomes: acceptability, adoption, appropriateness, feasibility, fidelity, costs, penetration and sustainability.
  Penetration: The integration of telemonitoring in the hospital. Assessment method by questionnaire.
Implementation outcome: Proctor Sustainability | Depending on each site and participant questionnaires are send out in 2025. Percentage: Whole study duration up untill the end of data analysis Feb 2028
  Implementation outcomes will be analyzed according to the taxonomy of Proctor et al. Proctor defined eight implementation outcomes: acceptability, adoption, appropriateness, feasibility, fidelity, costs, penetration and sustainability.
  Sustainability:The extent to which the use of telemonitoring is maintained within the hospital during and after the implementation phase. Assessment method: questionnaire and the percentage of centers that continued with telemonitoring after the implementation phase.

SECONDARY OUTCOMES:
Clinical outcome: All individual components of the primary, composite outcome | During pregnancy up to six months postpartum
Clinical outcome: Adverse perinatal event: Umbilical Cord Prolapse | During pregnancy and labour
Clinical outcome: Adverse perinatal event: Intrauterine infection requiring antibiotic treatment | During pregnancy up to six months postpartum
Clinical outcome: Healthcare consumption | During telemonitoring: average 11 days during pregnancy
  Number of days each participant received telemonitoring, as a proxy for the duration of in-hospital admission or outpatient visits potentially avoided. Additionally, number and indications of unplanned hospital visits and admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Depmann, Dr., Study Chair — UMC Utrecht
Locations (4):
- Netherlands (2):
  - Erasmus Medical Center Rotterdam (EMC), Rotterdam, South Holland
  - University Medical Center Utrecht (UMCU), Utrecht
- Catalan health institute: Vall d'Hebron University Hospital & Vall d'Hebron Research Institute (VHIR), Barcelona, Catalonia, Spain
- Region Stockholm: Karolinska Institutet, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bekker MN, Stephansson O, Maiz N, van der Kemp M, Ahaus K, Franx A. Digital healthcare as a solution for global challenges: A call for action. Acta Obstet Gynecol Scand. 2025 Feb;104(2):250-252. doi: 10.1111/aogs.15066. Epub 2025 Jan 28. No abstract available. PMID 39873168
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Bekker MN, Koster MPH, Keusters WR, Ganzevoort W, de Haan-Jebbink JM, Deurloo KL, Seeber L, van der Ham DP, Zuithoff NPA, Frederix GWJ, van den Heuvel JFM, Franx A. Home telemonitoring versus hospital care in complicated pregnancies in the Netherlands: a randomised, controlled non-inferiority trial (HoTeL). Lancet Digit Health. 2023 Mar;5(3):e116-e124. doi: 10.1016/S2589-7500(22)00231-X. PMID 36828605
- See also: European Perinatal Health Report: Core indicators of the health and care of pregnant women and babies in Europe from 2015 to 2019. — https://www.europeristat.com/publications/european-perinatal-health-report-2015-2019/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT07191236/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT07191236/ICF_001.pdf